CLINICAL TRIAL: NCT02936791
Title: Early PKD Observational Cohort Study
Acronym: EPOC
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00146013; U54DK126126 (NIH)
Record Dates: First submitted 2016-10-10; First posted 2016-10-18 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Polycystic Kidney Disease
Keywords: autosomal dominant polycystic kidney disease; ADPKD; PKD biomarkers; Kidney Institute; University of Kansas Medical Center
MeSH Terms: conditions — Polycystic Kidney Diseases; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood and urine samples are being collected from study participants. Researchers will only receive de-identified samples. No identifies will be given to investigators.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Individuals diagnosed with PKD: Individuals that have been diagnosed and meet the study's definition of early stage PKD.
- Individuals with a family history of PKD: Unaffected/ undiagnosed family members, preferably siblings, of participants with PKD
- Normal individuals for the comparison: Normal volunteers with no family history of PKD or other kidney diseases.

SUMMARY:
This observational study will collect blood and urine and clinical information from individuals with early-stages of polycystic kidney disease (PKD), their unaffected siblings and normal volunteers to create a biobank, also called a biorepository. The long-term goal is to develop new knowledge on biological markers or biomarkers that indicate changes in the disease progression. An understanding of biomarkers for early renal cyst growth will benefit PKD patients as new therapies are being developed and tested.

DETAILED DESCRIPTION:
In polycystic kidney disease (PKD), renal cysts form in utero and progressively enlarge due to aberrant proliferation of the cyst-lining cells and accumulation of fluid within the expanding cyst cavity. Over decades of unrelenting cyst growth, renal function declines due to the loss of functional tissue, eventually leading to kidney failure and the need for renal replacement therapy, such as dialysis or kidney transplantation.

Effective therapies for the treatment of PKD will need to be delivered as early as possible, before a measurable decline in kidney function, to preserve functional tissue. Currently, it is difficult to make an accurate prognosis of the progression of early-stage PKD since the growth of microscopic cysts is difficult to detect by standard imaging modalities and changes in total kidney volume measured within a reasonable time period are too small to be informative. Even though early cysts may not cause detectable changes in total kidney volume, their progressive enlargement damages the surrounding tissue and is a prelude to chronic kidney disease.

Current blood and urine tests provide important information on the decline of kidney function; however, these tests are not useful for monitoring early events of PKD such as initial cyst growth and damage to neighboring tissue. Clearly, novel biomarkers of early cystic disease need to be discovered to develop appropriate clinical tests to monitor the progression of early stage PKD. These tests will be important to identify patients at risk of rapid progression and of need of therapeutic intervention and to monitor the effectiveness of the therapeutic drug. The PKD Biomarkers Repository will allow approved researchers to obtain blood and urine samples for biomarker discovery and development of appropriate biomarker assays for prognosis of early PKD.

This observational study is currently recruiting for three groups: 1) individuals diagnosed with relatively early PKD as defined by total kidney volume and estimated GFR, 2) unaffected or undiagnosed family members, preferably siblings, 3) normal volunteers with no family history of renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion for early stage autosomal dominant polycystic kidney disease (ADPKD):

  * Family history of PKD
  * All races and ethnic groups
  * Glomerular filtration rate (GFR) >80 ml/min per 1.73 m2
* Inclusion for Healthy Volunteers:

  * Male or female with no family history of kidney disease
  * All races and ethnic groups
  * Normal GFR

Exclusion Criteria:

* Non-insulin or insulin-dependent diabetes mellitus
* Systemic illness (i.e.systemic lupus erythematosus, vasculitis)
* Unable to provide written informed consent
* Unavailable for magnetic resonance imaging (MRI) and blood/urine collection

Ages: 4 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The Study Population will include individuals clinically diagnosed with PKD and meet the inclusion criteria, their family members with not been diagnosed or have been determined not to have cysts within their kidneys and normal volunteers that will serve as a control group for the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Collect blood and urine samples from affected and unaffected cohorts for basic and translational research | 10 years
  The study will establish a repository of blood and urine from individuals with early stage PKD, unaffected/undiagnosed family members and normal volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Alan SL Yu, MD, Principal Investigator — University of Kansas Medical Center; Darren P Wallace, PhD, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PKD Biomarkers Repository Study — https://www.kumc.edu/research/kidney-institute/research/clinical-trials.html